CLINICAL TRIAL: NCT00278811
Title: Emergency Linkage to Outpatient Psychiatric Services
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Glenn Currier, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09541
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Emergency Services, Psychiatric
Keywords: Mental Health Services; Suicide; Suicide ideation
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: mobile crisis team

SUMMARY:
The purpose of this study is to compare two different kinds of follow-up care and their effects on psychiatric service use and psychological well-being. This randomized, controlled trial of subjects discharged from the psychiatric emergency services to outpatient care receive traditional hospital-based outpatient clinic referrals (treatment as usual) or appointments for community-based follow-up by a mobile crisis team.

DETAILED DESCRIPTION:
There are subgroups of patients who only seek care in emergency settings. An effective strategy to link that group to ambulatory care involves extending contact with psychiatric emergency services beyond the initial hospital-based visit. The "window of opportunity" to promote successful treatment linkage is brief. This is a study of a novel treatment format that seeks to expand the concept of the emergency contact, the study patients method of entering the mental health system of care, and by doing this, enhance retention in prescribed outpatient care. The effects of the intervention on patient symptoms and mental health service use will be examined.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish-speaking adult patients (18-and above) presenting to the psychiatric emergency service who rate a "1" or higher on the Spectrum of Suicidal Behavior of Pfeffer screening scale, and who have outpatient followup organized by Comprehensive Psychiatric Emergency Program staff through hospital outpatient psychiatric services are eligible for inclusion.

Exclusion Criteria:

* Subjects less than 18 years old, those rated as not suicidal in the emergency department, subjects with mental retardation/developmental delay, and subjects who have community psychiatric treatment that they elect to continue in lieu of hospital outpatient psychiatric services referral are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Subjects randomized to the experimental treatment will demonstrate significantly increased rates of linkage to first outpatient contact as compared with subjects randomized to control treatment. | 1 week

SECONDARY OUTCOMES:
Subjects randomized to experimental treatment will demonstrate significantly reduced levels of psychiatric symptoms and significantly increased scores of overall functioning at 3 months after study enrollment, | 3 months
and will demonstrate significantly higher use of outpatient mental health clinical services, lower use of ED contacts, and lower use of inpatient mental health services versus the control group during the six months after study enrollment. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenn W. Currier, M.D., M.P.H., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States